CLINICAL TRIAL: NCT02769637
Title: Effect of Acid Blockade on Microbiota and Inflammation in Cystic Fibrosis (CF)
Status: Terminated | Type: Observational
Why Stopped: unable to meet the target enrollment goal
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0672
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
Keywords: upper gastrointestinal tract; lung microbiota and inflammation
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA for 16S amplification
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ON PPI: Subjects on proton pump inhibitor (PPI) treatment
  Interventions: Drug: PPI treatment
- OFF PPI: Subjects off proton pump inhibitor (PPI) treatment

INTERVENTIONS:
Drug: PPI treatment — PPI treatment or no PPI treatment
  Other Names: Acid blockade medication
  Groups: ON PPI

SUMMARY:
Mucus in the airways of patients with CF represents an area for bacteria proliferation, microbial infection and inflammation. Similar to the lung, the esophagus provides an environment for bacterial to grow. The overall goal of this proposal is to characterize the esophageal microbiota of children with CF that are treated or untreated with acid blockade medication and to measure its possible impact on respiratory disease to develop novel treatment strategies.

DETAILED DESCRIPTION:
Patients with cystic fibrosis (CF) have significant morbidity and mortality due to airway infections. These infections are related to the deficiency of mucociliary clearance due to thick dehydrated secretions. Thus, considerable effort is spent managing airway infections. This includes therapies to improve mucus clearance and antibiotic treatments that target important pathogens. Understanding the source of airway microbiota, increased risk of infection, and exacerbation is critical to improve management of airway infection. A large proportion of CF patients are also treated with anti-acid medications. These medications decrease symptoms associated with gastroesophageal reflux disease (GERD), and improve the efficacy of enzyme replacement therapies. Critical for this proposal is the fact that aspiration may represent a potential route for airway infection from microorganisms in the upper gastrointestinal (GI) tract, and anti-acid treatments shift the GI microbiota. In preliminary studies we have identified a strong alteration of the esophageal microbiota in subjects using acid blocking medications. Thus, these treatments may have a significant effect on the bacterial communities present in the upper GI tract and may play a role in infection and exacerbation in CF. Traditionally, access to the upper GI tract has required endoscopy to acquire biopsy tissue, which is an invasive procedure and not routinely performed in CF. To circumvent the invasive sampling required for study of the esophagus we have recently shown that a minimally invasive test, the esophageal string test (EST), is capable of sampling the upper GI tract, and has performance comparable to biopsy for a number of measurements including assessment of the esophageal microbiota.

The primary hypothesis for this proposal is that acid blockade medication alters the esophageal microbiota in CF, increasing the presence of pathogenic bacteria and inflammation. To test this hypothesis we propose three Specific Aims:

Specific aim 1: Determine whether esophageal microbial composition in children with CF changes after withdrawal of acid blockade

1. Comparison of esophageal bacterial load by 16S qPCR in subjects on acid blockade and after withdrawal
2. Examine the stability of the esophageal bacterial communities based on longitudinal collection of the esophageal string test (EST) prior to withdrawal of acid blockade treatment.
3. Determine if there are changes after withdrawal of acid blockade in both sputum microbiota composition and esophageal microbiota (including presence of pathogenic bacteria) and whether the changes are correlated across the two sample types.

Specific aim 2: Determine whether esophageal microbiota in children with CF changes after initiation of acid blockade in patients started for clinical indications

1. Comparison of esophageal bacterial load by 16S qPCR of the esophageal bacteria in subjects pre and post acid blockade treatment.
2. Examine the stability of the esophageal bacterial communities based on longitudinal collection of the esophageal string test (EST) prior to acid blockade treatment initiation.
3. Determine if there are changes after initiation of acid blockade in both sputum microbiota composition and esophageal microbiota (including presence of pathogenic bacteria) and whether the changes are correlated across the two sample types.

Specific aim3: Examine the relation between acid blockade medication and inflammation in association with bacterial communities in subjects from aim 1 and 2

1. CompareIL-8 in the esophagus in subjects with and without acid blockade
2. Compare IL-8 in the sputum in subjects with and without acid blockade and determine relation between inflammation and association with shifts in the bacterial communities.

Together, these aims will provide novel information regarding the impact of acid blockade treatment on the esophageal and lung microbiota that may impact management of respiratory disease in CF. We anticipate similar effects of acid blockade on the esophageal bacterial communities as we observed in non-CF pediatric and adult subjects, but acknowledge that treatment burden in CF, particularly antibiotics, may affect the expected outcome. These data will provide critical information to evaluate the effect of acid blockade on infection risk, which could affect therapeutic choices for patients with CF. The long-term goal of these studies, is to improve patient care by assessing the effect of acid blocker therapy on the microbiota and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 10-21 years
2. Known diagnosis of CF based on sweat chloride > 60 mEq/L or identification of two known Cystic fibrosis transmembrane conductance regulator (CFTR) mutations
3. Clinically stable pulmonary disease defined by

   1. clinical impression of patient's primary CF provider,
   2. no newly prescribed antibiotic treatments in the 30 days prior to enrollment, and
   3. relativly stable lung function with a forced expiratory volume in 1 second (FEV1) within 10% of baseline.
4. Male and female
5. Willing to participate in and comply with all study procedures, and
6. Willingness of the subject, parent or legally authorized representative to provide written informed consent.
7. Body Mass Index (BMI) >25%
8. >40% FEV1.
9. Willing to stop acid blockade medication for 6 weeks for aim 1.
10. Not on acid blockade for 6 weeks for aim 2.

Exclusion Criteria:

1. FEV1 less than 40% predicted
2. History of meconium ileus, distal intestinal obstructive syndrome, gastrointestinal surgery, or intestinal stricture.
3. CF liver disease with cirrhosis, gastric or esophageal varices.
4. Unwilling to participate in and comply with the study procedures.
5. Unwillingness of the subject, parent or legally authorized representative to provide written informed consent.
6. Unwilling or unable to swallow the capsule with the esophageal string test (EST).
7. Gelatin allergy.
8. History of esophageal surgery including fundoplication, or
9. Presence of a gastrostomy tube.
10. Confirmed or suspected diagnosis of Gastroesophageal Reflux Disease (GERD)
11. BMI < 25%

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with Cystic Fibrosis
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Changes in the microbiota and inflammation | Baseline and 6 weeks
  Identification of bacterial communities and IL-8

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Fillon, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No